CLINICAL TRIAL: NCT05430035
Title: Safety and Feasibility of Prophylactic Heated Intra-peritoneal Chemotherapy (HIPEC) for High-Risk Gallbladder Adenocarcinoma
Brief Title: Safety and Feasibility of HIPEC for High-Risk Gallbladder Adenocarcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Brian Boone, MD, FACS, Assistant Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2202522011
Record Dates: First submitted 2022-06-17; First posted 2022-06-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Gallbladder Adenocarcinoma
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HIPEC (Experimental): Prophylactic Heated Intra-peritoneal Chemotherapy (HIPEC) 30 mg of mitomycin C (MMC) over the first 60 minutes followed by 10 mg over an additional 30 minutes. Perfusate will be heated to obtain a tissue temperature of 42°.
  Interventions: Drug: HIPEC

INTERVENTIONS:
Drug: HIPEC — Heated Intra-Peritoneal Chemotherapy (HIPEC) HIPEC will be performed at the time of the index operation if a cancer is known pre-operatively, at the time of re-operation for incidentally discovered cancers already treated with cholecystectomy that are undergoing central hepatectomy and portal lymphadenectomy as part of standard of care, or independently if no other procedures are indicated. A closed technique will be utilized to deliver mitomycin C (MMC) over the first 60 minutes followed by an additional smaller dose over an additional 30 minutes. Perfusate will be heated to obtain a tissue temperature of 42°
  Other Names: intra-peritoneal chemotherapy; mitomycin c

SUMMARY:
Gallbladder adenocarcinoma is a devastating disease associated with a poor prognosis. Gallbladder and other biliary cancers will be responsible for an estimated 11,980 new cases, and 4,090 deaths in the US during 2020. The 5-year survival for all patients with gallbladder cancer is 18%, however this plummets to 2% for patients with metastatic disease. Patients with gallbladder cancer frequently develop peritoneal recurrence, particularly after intra-operative bile spillage during cholecystectomy for incidentally discovered gallbladder malignancy. Once developed, peritoneal metastases are difficult to treat and result in significant morbidity and mortality. As a result, novel approaches that target peritoneal metastases are needed for this disease. Prophylactic use of heated intraperitoneal chemotherapy (HIPEC) has been explored or is under active investigation for numerous gastrointestinal malignancies, including colon, gastric, and appendiceal cancers. HIPEC has efficacy in gallbladder cancer patients with macroscopic peritoneal disease undergoing cytoreductive surgery (CRS)/HIPEC and has been associated with a survival advantage in a multi-institutional retrospective case series. Incidentally discovered gallbladder cancer is treated with central hepatectomy and portal lymphadenectomy, therefore a prophylactic HIPEC can be easily incorporated into the second operation performed as part of the standard of care. In this early phase clinical trial, the investigators will explore the safety and feasibility of prophylactic HIPEC for gallbladder cancer in patients at high-risk of peritoneal recurrence. The primary endpoint is to assess feasibility of the prophylactic heated intraperitoneal chemotherapy (HIPEC) approach in gallbladder cancer. The primary endpoints include occurrence of intra-operative complications, technical challenges, 90-day postoperative morbidity and mortality, length of stay and readmission, which will be documented and compared with historical controls after follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed gallbladder adenocarcinoma AND inadvertent spillage of bile or intentional decompression during cholecystectomy OR tumors extending through the serosa of the gallbladder (T3/T4) OR poorly differentiated gallbladder adenocarcinoma.
* ECOG Performance status ≤ 2
* Subjects must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 10.0 g/dl
  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine within normal institutional limits
* Eligible TNM staging includes >T1b meeting above criteria, any N, and M0
* Eligible candidates for standard surgical management which includes central liver resection (+ cholecystectomy if not already performed) and portal lymphadenectomy
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior systemic therapy for gallbladder adenocarcinoma
* Subjects receiving any other investigational agents.
* Subjects with known or suspected metastatic disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MMC or other agents used in this study.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding are excluded from this study because MMC has the potential for teratogenic or abortifacient effects. Because there is known risk for adverse events in nursing infants secondary to treatment of the mother with MMC, breastfeeding should be discontinued if the mother is treated with MMC.
* Subjects with past medical history of hepatitis B or C
* Subjects with evidence of biliary obstruction thought to be cancer related, including subjects requiring biliary stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Occurrences of intraoperative complications | During procedure
  Number of occurrences of intraoperative complications
Occurrences of Postoperative Morbidity and Mortality | 90 days postoperative
  Number of occurrences of postoperative morbidity and mortality
Length of Stay | Up to 90 days
  LOS Median
Readmission | Up to 90 days
  Number of readmission occurrences

SECONDARY OUTCOMES:
Peritoneal Metastases | Up to 5 Years
  Incidence of Peritoneal Metastases
Disease Free Survival | Up to 5 Years
  Incidence of Disease Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Brian Boone, MD, Principal Investigator — WVU Cancer Institute
Locations (1):
- West Virginia University Cancer Institute Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States